CLINICAL TRIAL: NCT02273089
Title: Use of CPAP to Reduce Arterial Stiffness in Moderate to Severe Obstructive Sleep Apnea, Without Excessive Daytime Sleepiness (STIFFSLEEP)
Brief Title: CPAP to Reduce Arterial Stiffness in Non Sleepy, Moderate to Severe Obstructive Sleep Apnea (STIFFSLEEP)
Acronym: STIFFSLEEP
Status: Terminated | Type: Observational
Why Stopped: Recruitment stopped due to time restrains
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: CHLC.CI.105.2014
Record Dates: First submitted 2014-10-06; First posted 2014-10-23 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Obstructive Sleep Apnea; Vascular Stiffness; Sleep Disorder Daytime Somnolence
Keywords: Obstructive sleep apnea; arterial stiffness; CPAP; excessive daytime sleepiness; pulse wave velocity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disorders of Excessive Somnolence | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- OSA w/o EDS: Males with moderate to severe obstructive sleep apnea without excessive daytime sleepiness will be proposed nocturnal CPAP (ResMed S9 AutoSet) for three months
  Interventions: Device: CPAP (ResMed S9 AutoSet)
- OSA w EDS: Males with moderate to severe obstructive sleep apnea with excessive daytime sleepiness will be proposed nocturnal CPAP (ResMed S9 AutoSet) for three months
  Interventions: Device: CPAP (ResMed S9 AutoSet)

INTERVENTIONS:
Device: CPAP (ResMed S9 AutoSet) — nocturnal CPAP for three months

SUMMARY:
This study intends to determine whether continuous positive airway pressure (CPAP) can reduce arterial stiffness (measured by pulse wave velocity) in nonsleepy as well as in sleepy patients with obstructive sleep apnea .

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is associated with increased cardiovascular morbidity and mortality. Arterial stiffness, evaluated by pulse wave velocity, is related to atherosclerosis and cardiovascular risk. It has been reported that arterial stiffness is higher in patients with OSA than in healthy control groups, and it is assumed that it decreases after treatment with CPAP.

In patients with OSA without daytime hypersomnolence it is not clear if CPAP has some benefits on cardiovascular events and hypertension.

This study aims to evaluate the effect of CPAP therapy in an interventional cohort of patients with moderate to severe OSA, in which each patient will be is own control, for ethical reasons; the effect of CPAP therapy on the subcohorts of sleepy and of nonsleepy patients will be compared. The effect of a three months trial of CPAP will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe obstructive sleep apnea, defined as apnea/hypopnea index superior to 15

Exclusion Criteria:

* Epworth sleep scale superior to 16
* other sleep diseases
* moderate or severe lung disease
* cardiac disease other than hypertension
* cerebrovascular diseases
* other vascular diseases
* other chronic diseases except metabolic syndrome

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with moderate to severe obstructive sleep apnea, with or without excessive daytime sleepiness
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Aortic pulse wave velocity (PWV) | Change on PWV from baseline up to three months of intervention
  carotid-femoral (aortic) pulse wave velocity (PWV) measured by noninvasive piezo-electronic system with Complior(R) (Colson, France).

SECONDARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | Change on AHI from baseline up to three months of intervention
  AHI is an index used to assess the severity of sleep apnea based on the total number of complete cessations (apnea) and partial obstructions (hypopnea) of breathing occurring per hour of sleep, using polygraphic study.
Nocturnal oxygenation | Change from baseline up to three months of intervention
  Measure of minimal saturation of oxygen (SO2), time under 90% SO2, average SO2, oxygen desaturation index, using polygraphic study.
Excessive daytime sleepiness | Change on ESS from baseline up to three months of intervention
  Epworth sleep scale (ESS)

OTHER OUTCOMES:
Lipidic profile | Change from baseline up to three months of intervention
  total serum cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides
Glucidic profile | Change from baseline up to three months of intervention
  fasting serum glucose and HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Mineiro, MD, Principal Investigator — Centro Hospitalar de Lisboa Central; Pedro Marques-da-Silva, MD, Study Chair — Centro Hospitalar de Lisboa Central; João Cardoso, MD, Study Chair — Centro Hospitalar de Lisboa Central; Maria João Marques-Gomes, MD, PhD, Study Director — Universidade Nova de Lisboa
Locations (2):
- Portugal (2):
  - Consulta de Sono, Departamento de Pneumologia, Centro Hospitalar de Lisboa Central, Lisbon
  - Núcleo de Hipertensão Arterial, Consulta de Medicina do Hospital de Santa Marta, Centro Hospitalar de Lisboa Central, Lisbon

REFERENCES:
- [Derived] Mineiro MA, Silva PMD, Alves M, Papoila AL, Marques Gomes MJ, Cardoso J. The role of sleepiness on arterial stiffness improvement after CPAP therapy in males with obstructive sleep apnea: a prospective cohort study. BMC Pulm Med. 2017 Dec 8;17(1):182. doi: 10.1186/s12890-017-0518-z. PMID 29221483
- [Derived] Mineiro MA, Marques da Silva P, Alves M, Virella D, Marques Gomes MJ, Cardoso J. Use of CPAP to reduce arterial stiffness in moderate-to-severe obstructive sleep apnoea, without excessive daytime sleepiness (STIFFSLEEP): an observational cohort study protocol. BMJ Open. 2016 Jul 12;6(7):e011385. doi: 10.1136/bmjopen-2016-011385. PMID 27406645